CLINICAL TRIAL: NCT04250896
Title: Using Behavioral Science and mHealth Tools for Early Prevention of Childhood Obesity in Mexico
Brief Title: mHealth for Prevention of Childhood Obesity in Mexico
Acronym: mHealth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mexican National Institute of Public Health (Other Government)
Collaborators: UNICEF (Other)
Responsible Party: Principal Investigator, Anabelle Bonvecchio Arenas, Director of Research in Nutrition Policies and Programs, Mexican National Institute of Public Health
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: CI1547
Record Dates: First submitted 2019-10-31; First posted 2020-01-31 (Actual); Last update posted 2021-09-14 (Actual); Status verified 2021-09

CONDITIONS: Overweight and Obesity
Keywords: Randomised controlled trial; Text messaging; Infant feeding practice; health unit; BMI; Mobile phone; prevention
MeSH Terms: conditions — Overweight; Obesity | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: Control group will receive standard child care in health units plus exposure to EsIAN (Strategy of Integral Attention to Nutrition of Mexico). At the same time as the intervention group, in addition to the control group, will receive SMS through a cell pone on practices related to the prevention of infant malnutrition (in primary caregivers) and the strengthening of counseling for the prevention of infant malnutrition with health providers.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: The randomized unit is the health center
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Other): Control group will receive standard child care in health units plus exposure to EsIAN (Strategy of Integral Attention to Nutrition)
  Interventions: Other: Control group
- Intervention (Experimental): Intervention group will receive SMS messages sent through a cell pone in addition to the control group receive (standard child care in health units plus exposure to EsIAN)
  Interventions: Behavioral: SMS´s sending by cell phone for behavior change

INTERVENTIONS:
Other: Control group — Standard child care in health unit plus exposure to EsIAN
  Arms: Control
Behavioral: SMS´s sending by cell phone for behavior change — SMS messages sent through a cell pone through the RapidPro platform on practices related to the prevention of infant malnutrition to primary caregivers and the strengthening of counseling for the prevention of infant malnutrition with health providers.
  Arms: Intervention

SUMMARY:
Background: The sending of text messages (short messaging service, SMS) has been proven as an effective strategy in behavior change. In Mexico, the Strategy of Comprehensive Care for the Nutrition (EsIAN for its acronym in Spanish ) focuses on improving access to information for the main caregivers of child beneficiaries on the practice of infant feeding and healthy physical activity.

Objective: To assess whether the mHealth (or mobile health) strategy or the sending of SMS has an effect on knowledge, attitudes, intentionality, perceived control and practices to prevent childhood malnutrition in a population living in poverty.

Design: Randomized effectiveness trial by conglomerates. Participants: 400 primary caregivers of children <59 months and health personnel working in the health units included in the study.

Control group: Healthy child care in standard health units plus exposure to EsIAN.

Intervention group: In addition to the control group, the SMS are sent through a cell pone through the RapidPro platform on practices related to prevention of child malnutrition (in primary caregivers) and the reinforcement of counseling for the prevention of infant malnutrition (with health personnel).

Randomization: The first level health units were stratified by state (Morelos or Yucatan); rural and urban area and affiliation institution (Secretary of Health or Mexican Institute of Social Security); and randomized to be assigned to the control or intervention group; 400 primary caregivers of children <59 months in total will be included for the study.

Main measures of interest: State of nutrition and knowledge, attitudes or practices on breastfeeding, physical activity, adoption and preparation of healthy foods and beverages in primary caregivers of children<5 years old; and advice on the key messages of EsIAN by health providers.

DETAILED DESCRIPTION:
RapidPro is a tecnological platform of programming of short messaging service (SMS) for cell phone.

Morelos is the name of one of the central states of Mexico Yucatan is the name of one of the south states of Mexico

ELIGIBILITY:
Inclusion Criteria:

* Primary caregivers whose beneficiaries children are cared in the health units selected for the study and who have a cell pone in home
* Health personnel who provides services to Prospera population in the health units selected for the study and that have a cell pone
* Primary caregiver, must care for at least one child under 60 months users of the health units selected for the study

Exclusion Criteria:

* Primary caregivers and health personnel who do not have a cell pone or who do not have connectivity in their communities
* Health personnel, who have been in office for a least 3 months

Max Age: 59 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1000 (Actual)
Dates: Start 2020-08-01 (Actual); Primary Completion 2020-11-01 (Actual); Study Completion 2021-09-06 (Actual)

PRIMARY OUTCOMES:
prevalence of overweight and obesity | basal and through study completion, an average of 9 months.
  Through the measurements of weight and height to children under 60 months, the estimator of body mass index adjusted for age will be calculated to determine prevalence of overweight (+1 SD. Z score ) and obesity (+2 SD Z score).

SECONDARY OUTCOMES:
Proportion of caregivers / mothers with correct infant feeding practices scale | basal and through study completion, an average of 9 months.
  Practices related to breastfeeding, complementary food and healthy nutrition during childhood (scale of 0-20 values , which high scores >15 is correct)
Proportion of caregivers / mothers with correct physical activity practices scale | basal and through study completion, an average of 9 months.
  Practices of physical activity to less 5 years old (scale of 0-20 values , which high scores >15 is correct)

OTHER OUTCOMES:
knowledge and attitudes related to infant feeding practices and physical activity of child | basal and through study completion, an average of 9 months.
  scales of knowledge and attitudes about nutrition and physical activity of the child (scale of 0-5 values, which high scores is agreement or very important)

CONTACTS AND LOCATIONS:
Overall Officials: Anabelle Bonvecchio, PhD, Principal Investigator — Mexican National Institute of Public Health
Locations (1):
- Ministry of Health of Morelos State, Cuernavaca, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lozada-Tequeanes AL, Theodore FL, Kim-Herrera E, Garcia-Guerra A, Quezada-Sanchez AD, Alvarado-Casas R, Bonvecchio A. Effectiveness and Implementation of a Text Messaging mHealth Intervention to Prevent Childhood Obesity in Mexico in the COVID-19 Context: Mixed Methods Study. JMIR Mhealth Uhealth. 2024 Apr 9;12:e55509. doi: 10.2196/55509. PMID 38592753